CLINICAL TRIAL: NCT03077815
Title: National Taiwan University Hospital
Brief Title: Systematically Intermittent Arm Exercise for Improving Maturation of Hemodialysis Arteriovenous Shunt: Study Protocol for a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201701043RINC
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2018-12

CONDITIONS: Systematically Intermittent Arm Exercise for Improving Maturation of Hemodialysis Arteriovenous Shunt

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm movement more than a total of at least 30 minutes a day (Other): Using the provided rubber ball grip the ball movement on a daily basis, and grip the ball at a time 3-5 seconds, every 5 minutes, daily at least 6 rounds (for example, according to the daily morning, noon and night-time sports training in the two groups), to reach an arm movement more than a total of at least 30 minutes a day
  Interventions: Other: Systematically intermittent arm exercise
- arm movement and local press strength 50 mmHg at the upper arm (Other): Using the provided rubber ball grip the ball movement on a daily basis, and grip the ball at a time 3-5 seconds, every 5 minutes, daily at least 6 rounds (for example, according to the daily morning, noon and night-time sports training in the two groups), to reach an arm movement more than a total of at least 30 minutes a day with Elbow proximal 4 (2~6) local press strength 50 mmHg at the upper arm
  Interventions: Other: Systematically intermittent arm exercise

INTERVENTIONS:
Other: Systematically intermittent arm exercise — While holding a rubber ball for 5 minutes a day, together with strappy elastic compression arm veinElastic bandages defined for using this research provides of standard bandages, according to research personnel Guide, reached hand elbow near heart end 4 (2~6) cm at of arm local pressure strong 50 mm-Hg (+/-10 mm-Hg) (about equivalent to provides pressure strong 6.67 thousand PA (kPa), also about equivalent to 0.97 PSI (pound per square inch)), to reached 5 minutes arm movement Shi short reduced vein return, promotion pathway vein extended of effect
  Other Names: Systematically intermittent arm exercise with local pressure

SUMMARY:
Arm vein intermittently gripping arm movements, can promote the increased diameter of arteriovenous fistula, which enhance the maturity of fistula, the effect of lack of empirical research. Objective: this study, randomized controlled study, investigate systematic random arm vein pressure and arm movements to arteriovenous fistula in hemodialysis patients improve the maturity rate and effectiveness of the diameter. Methods: a prospective comparative study randomly assigned.

DETAILED DESCRIPTION:
the effect size is the diameter of arteriovenous fistula in hemodialysis patients with treatments or not is the key to smoothly. Arm vein intermittently gripping arm movements, can promote the increased diameter of arteriovenous fistula, which enhance the maturity of fistula, the effect of lack of empirical research. Objective: this study, randomized controlled study, investigate systematic random arm vein pressure and arm movements to arteriovenous fistula in hemodialysis patients improve the maturity rate and effectiveness of the diameter. Methods: a prospective comparative study randomly assigned. This study plan for each patient has received a wrist artery and vein access tracks before and after 3 months of operation, according to randomly divided into three groups, the first group of patients after accepted guidance for systematic and intermittent arm movements; the second group of patients receiving the guidance system of intermittent arm vein compression and arm movements; a third group as a control group. Discussion: the plan is expected to include 150 patients, receive instruction after the randomly with/without systemic venous pressure, with/without systemic movement. The plan design under the patient safety assessment of the effectiveness of these two activities the primary end point and secondary end points. This study offers clinicians advise patients, how to effectively improve the patients ' arteriovenous access matured speed and diameter. Keywords: Arteriovenous shunt, compression bandages, exercise therapy, renal dialysis

ELIGIBILITY:
Inclusion Criteria:

* Inclusion for adult patients aged 20 and above. Preoperative evaluation site assessment/operation condition full wrist wrist artery and vein arteriovenous joint surgery. Objective sufficient conditions are defined as wrist artery and vein,/objective ultrasound evaluation before surgery, vein of the arm extended diameter scan before >= 2.5 mm, radial natural >= 2.0 mm diameter scan, no significant narrowing of both forearm. Excluded conditions including following, joined research Qian found patients too weak/or heart failure too serious/or consciousness not clear/or long-term bed, both inside and outside section attending operation Qian excluded wrist Department moving vein pathway surgery; operation Qian assessment/surgery site assessment wrist Department moving vein conditions insufficient, surgery physician judge to for standard wrist Department moving vein pathway/or select standard junction bit yiwai of parts for surgery; surgery Shi occurred non-expected negative complications, cannot effective completed surgery And said it could not meet before joining the research or patient tracking movement refused to examine the test or measurement

Exclusion Criteria:

* weak / serious heart failure / unclear / long-term bed rest, internal and external surgery physician preoperative removal of wrist arteriovenous access surgery; preoperative assessment / surgery site evaluation of wrist arteriovenous conditions, the surgeon to determine The standard wrist arteriovenous access and / or the selection of part of the standard joint site for surgery; unintended adverse complications during surgery, can not effectively complete the surgery; within one week after surgery complications, not suitable for tracking exercise or measurement, or before the study The patient indicated that he could not cooperate with the tracking exercise or the measurement and refused to study the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 119 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The diameter of each passage of the passage vein (forearm head vein) of the arterial and venous access within three months | Postoperative Three months
  Comparison of the various methods to achieve within three months the checkpoint path diameter increase rate (two time points measurement difference).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Chan, phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, No.7, Chung Shan S. Rd, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JW, Fu HY, Hii IH, Tseng HW, Chang PY, Chang CH, Chen YS, Hsu RB, Wu IH, Chen YM, Chu TS, Hung KY, Lin SL, Wu KD, Chan CY. A Randomized Trial of Postoperative Handgrip Exercises for Fistula Maturation in Patients With Newly Created Wrist Radiocephalic Arteriovenous Fistulas. Kidney Int Rep. 2022 Dec 24;8(3):566-574. doi: 10.1016/j.ekir.2022.12.019. eCollection 2023 Mar. PMID 36938082